CLINICAL TRIAL: NCT02109458
Title: Navigational Bronchoscopy and Transthoracic Needle Biopsy for the Diagnosis of Peripheral Pulmonary Nodules: A Safety and Feasibility Pilot
Brief Title: Pilot Study of Navigational Bronchoscopy and Transthoracic Needle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Veran Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00086035
Record Dates: First submitted 2014-03-17; First posted 2014-04-10 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Peripheral Pulmonary Nodules
Keywords: Lung nodule biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assessing peripheral pulmonary nodules (Experimental): To evaluate the feasibility and safety of a procedure path including convex Endobronchial Ultrasound (EBUS) lymph node sampling, navigation guided bronchoscopy (NB) and navigation guided transthoracic needle aspiration (N-TTNA).
  Interventions: Device: Navigation guided bronchoscopy

INTERVENTIONS:
Device: Navigation guided bronchoscopy — Navigation guided transthoracic needle aspiration (N-TTNA) and navigation guided bronchoscopy (NB); guidance system is by Veran Medical Technologies, Inc.

SUMMARY:
The goal of this study is to evaluate the feasibility and safety of navigation guided virtual transthoracic needle biopsy combined with navigational bronchoscopy for the diagnosis of peripheral pulmonary nodules (PPN).

DETAILED DESCRIPTION:
Accessing peripheral pulmonary nodules is problematic because they are often not visible endobronchially, not large enough to be visualized by x-ray fluoroscopy for transbronchial biopsy (TBBx), and/or do not lie within an accessible airway. In this study, investigators hope to evaluate new technologies to aid in PPN biopsy using navigation bronchoscopy (NB) combined with navigation transthoracic needle aspiration (N-TTNA) sampling of a PPN.

Patients meeting inclusion criteria who consent will undergo a convex Endobronchial Ultrasound (EBUS) bronchoscopy for evaluation and sampling of the mediastinum and hilum. Following this, NB will be performed with an ultrathin bronchoscope (4mm outer diameter with a 2 mm working channel) with R-EBUS and fluoroscopy. If the lesion is localized by NB and/or radial EBUS in conjunction with NB, TBBX will be taken. At the conclusion of TBBX sampling, a fluoroscopic evaluation to assess for the presence of pneumothorax will be performed and if one is present, appropriate clinical measures will be taken at the discretion of the treating team (tube thoracostomy, observation, etc.) and no further sampling techniques will be utilized. If the lesion was not able to be localized via NB and/or the physician feels insufficient sample was acquired for diagnosis and there is no evidence of pneumothorax, the patient will undergo N-TTNA at the same PPN during the same procedure time. It is envisioned that between 8-12 patients will require a N-TTNA to complete diagnosis.

ELIGIBILITY:
Inclusion criteria:

* Target patient population: Patients with a peripheral pulmonary nodule as identified on CT chest ≤3cm from the pleura will be recruited. A PPN will be defined as a lesion >10mm and <3cm in diameter surrounded by lung parenchyma on CT chest. The decision for biopsy of the PPN will be made by the treating physician and agreed upon by the patient.
* Participants must be at least 18 years old or older
* No bleeding disorders
* Provide informed consent.

Exclusion criteria

* less than 18 years
* lack of fitness for flexible bronchoscopy as determined by the physician performing the bronchoscopy before the procedure
* inability to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Assessing Peripheral Pulmonary Nodules: To evaluate the feasibility and safety of a procedure path including convex Endobronchial Ultrasound (EBUS) lymph node sampling, navigation guided bronchoscopy (NB) and navigation guided transthoracic needle aspiration (N-TTNA).
  Navigation guided bronchoscopy
Period: Overall Study
Arm/Group | Assessing Peripheral Pulmonary Nodules
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Assessing Peripheral Pulmonary Nodules: To evaluate the feasibility and safety of a procedure path including convex EBUS lymph node sampling, navigation guided bronchoscopy (NB) and navigation guided transthoracic needle aspiration (N-TTNA).
  Navigation guided bronchoscopy
Arm/Group | Assessing Peripheral Pulmonary Nodules
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: Feasibility assessed by number of participants with successful completion of biopsy (i.e. a biopsy was able to be obtained to collect a tissue sample)
Time Frame: Immediately following procedure
Measure: Number; unit: participants
Arm/Group | Assessing Peripheral Pulmonary Nodules
Number analyzed (Participants) | 24
participants | 24

2. Primary Outcome: Incidence of Pneumothorax
Description: Presence of pneumothorax assessed in participants with successful completion of biopsy.
Time Frame: Immediately after procedure
Measure: Number; unit: participants
Arm/Group | Assessing Peripheral Pulmonary Nodules
Number analyzed (Participants) | 24
participants | 5

3. Secondary Outcome: Positive Diagnostic Yield of Bronchoscopic Biopsy of Electromagnetic Guidance Trans-thoracic Needle Aspiration (ETTNA) Alone
Description: Positive diagnostic yield of bronchoscopic biopsy of Electromagnetic Guidance Trans-thoracic Needle Aspiration (ETTNA) alone was defined by participants having benign or malignant pathology.
Time Frame: Approximately 1 week upon receipt of pathology report
Measure: Number; unit: participants
Arm/Group | Assessing Peripheral Pulmonary Nodules
Number analyzed (Participants) | 24
participants | 19

4. Secondary Outcome: Positive Diagnostic Yield of Bronchoscopic Biopsy of ETTNA + EBUS + NB
Description: Positive diagnostic yield of bronchoscopic biopsy of ETTNA + EBUS + NB was defined by participants having benign or malignant pathology.
Time Frame: Approximately 1 week upon receipt of pathology report
Measure: Number; unit: participants
Arm/Group | Assessing Peripheral Pulmonary Nodules
Number analyzed (Participants) | 24
participants | 21

ADVERSE EVENTS:
Arm/Group | Assessing Peripheral Pulmonary Nodules
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assessing Peripheral Pulmonary Nodules (N=24)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) — Blood in sputum

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes